CLINICAL TRIAL: NCT04227912
Title: Comparison of Postoperative Analgesic Efficacy of Preemptive Ultrasound-guided Transversus Abdominis Plane Block, Ultrasound-guided Local Infiltration and Intravenous Dexketoprofen in Inguinal Hernia Repair
Brief Title: Transversus Abdominis Plane(TAP) Block, Local Infiltration and Intravenous Dexketoprofen in Inguinal Hernia Repair
Acronym: Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fikret Salık, Assistant Professor, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SBUGaziYasargilTRH
Record Dates: First submitted 2020-01-08; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group TAP (Active Comparator): Ultrasound-guided TAP Block
  Interventions: Other: Transversus abdominis plane block
- Group Local (Active Comparator): Ultrasound-guided Local Infiltration
  Interventions: Other: Local anesthetic infiltration
- Group Dexketoprofen (Active Comparator): Intravenous Dexketoprofen
  Interventions: Other: Intravenous dexketoprofen

INTERVENTIONS:
Other: Transversus abdominis plane block — Before surgery, Ultrasound-guided TAP block was performed preemptively to Group TAP patients.
  Arms: Group TAP
Other: Local anesthetic infiltration — Before surgery, Ultrasound-guided Local anesthetic infiltration to the surgical incision line was performed preemptively to Group Local patients.
  Arms: Group Local
Other: Intravenous dexketoprofen — Before surgery, 50 mg intravenous dexketoprofen was performed preemptively to Group dexketoprofen patients.
  Arms: Group Dexketoprofen

SUMMARY:
This study evaluates the compare the effects of ultrasound guided TAP block, local anesthetic infiltration to the incision line and intravenous dexketoprofen on postoperative analgesic efficacy and rescue tramadol consumption in inguinal hernia repairs.

DETAILED DESCRIPTION:
Currently, multimodal techniques are used in inguinal hernia repairs in addition to pharmacological and regional techniques for postoperative analgesia.TAP block is performed on the principle of hydrodissection of the fascia between the internal oblique and transversus abdominis muscles of the abdominal wall muscles with local anesthetic drugs. Local anesthetic drugs provide analgesic effect up to 24 hours in the postoperative period by blocking the T6-L1 nerves in the facial plane. Local anesthetic infiltration which is one of the regional anesthetic techniques, is another method of postoperative analgesia. intravenous analgesic drug is also used as pharmacological postoperative analgesia method in most clinics.

ELIGIBILITY:
Inclusion Criteria:

* Subject who aged 18-75 years
* American Society of Anesthesiologist (ASA) I-III
* Subject undergoing unilateral or bilateral inguinal hernia repair

Exclusion Criteria:

* Subject under 18 and over 75 years of age
* ASA IV
* History of allergy to agents
* Analgesic drug use in the last 48 hours
* Morbid obese (BMI> 35)
* Confusion
* Coagulopathy
* Local infection at the injection site
* Subject with heart, lung, hematologic, metabolic and endocrine disease
* Subject who did not want to be included in the study
* Subject who refused the spinal anesthesia
* Subject who failed the spinal anesthesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Postoperative rescue tramadol consumption | 24 hours
  The mean tramadol consumption in the first 24 post-operative hours

SECONDARY OUTCOMES:
Analgesic efficacy | 24 hours
  Postoperative visual analog scale score recorded 0-10 (0 = no pain, 10 = severe pain) at 30. min, 1, 2, 4, 8, 12, 16 and 24 hours postoperatively
Postoperative nausea-vomiting | 24 hours
  Postoperative nausea-vomiting was evaluated with a 3-point system (0: no nausea and vomiting, 1: nausea, but no vomiting, 2: nausea with or without nausea) 24 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Fikret Salık, Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Locations (1):
- University of Health Sciences Gazi Yaşargil Training and Research Hospital, Diyarbakır, Eyalet/Yerleşke, Turkey (Türkiye)

REFERENCES:
- [Result] Joshi GP, Rawal N, Kehlet H; PROSPECT collaboration; Bonnet F, Camu F, Fischer HB, Neugebauer EA, Schug SA, Simanski CJ. Evidence-based management of postoperative pain in adults undergoing open inguinal hernia surgery. Br J Surg. 2012 Feb;99(2):168-85. doi: 10.1002/bjs.7660. Epub 2011 Sep 16. PMID 21928388
- [Result] Petersen PL, Mathiesen O, Stjernholm P, Kristiansen VB, Torup H, Hansen EG, Mitchell AU, Moeller A, Rosenberg J, Dahl JB. The effect of transversus abdominis plane block or local anaesthetic infiltration in inguinal hernia repair: a randomised clinical trial. Eur J Anaesthesiol. 2013 Jul;30(7):415-21. doi: 10.1097/EJA.0b013e32835fc86f. PMID 23549122
- See also: European Journal of Anaesthesiology — https://insights.ovid.com/